CLINICAL TRIAL: NCT05548933
Title: Effects of Nonsurgical Periodontal Therapy on Biomarkers in Serum and Gingival Crevicular Fluid in Severe Periodontitis (Stage III/IV) and Hyperlipidemia:A Cohort Study
Brief Title: Effects of Non-surgical Periodontal Therapy on Severe Periodontitis and Hyperlipidemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0567
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Periodontitis Chronic Generalized Severe; Hyperlipidemia; Gingival Crevicular Fluid; Serum; Biomarkers; Non-surgical Periodontal Therapy
Keywords: severe periodontitis; hyperlipidemia; gingival crevicular fluid; serum; biomarkers; non-surgical periodontal therapy
MeSH Terms: conditions — Hyperlipidemias; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HP: Chronic periodontitis (stage III/IV) patients with hyperlipidemia
  Interventions: Procedure: non-surgical periodontal therapy
- CP: Chronic periodontitis(stage III/IV) patients without hyperlipidemia
  Interventions: Procedure: non-surgical periodontal therapy

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — supragingival scaling,subgingival scaling

SUMMARY:
This study was a single-center, non-randomized, parallel-group design clinical trial, and each group was assigned a 1:1 ratio with or without hyperlipidemia. Both groups underwent periodontal non-surgical treatment, and blood and gingival crevicular fluid were collected before surgery, 1 month and 3 months after surgery for the detection of MCP-1, IL-8, oxLDL, TNF-α, TG, LDL-C, HDL-C.

DETAILED DESCRIPTION:
This study was a single-center, non-randomized, parallel-group design clinical trial, and each group was assigned a 1:1 ratio with or without hyperlipidemia. Both groups underwent periodontal non-surgical treatment, and blood and gingival crevicular fluid were collected before surgery, 1 month and 3 months after surgery for the detection of MCP-1, IL-8, oxLDL, TNF-α, TG, LDL-C, HDL-C.MCP-1, IL-8, oxLDL, TNF-α will be tested for concentration using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to meet at least one of the following criteria for the diagnosis of hyperlipidemia: triglyceride (TRG) levels >2.26 mmol/L; high density lipoprotein cholesterol (HDL-C) levels <1.04 mmol/L; or low density lipoprotein cholesterol (LDL-C) levels >4.14 mmol/L
* Patients with severe periodontitis (stage III/IV) with probing depth (PD) ≥ 6 mm at at least six sites, at least two multi-rooted or two single-rooted teeth in at least one quadrant, and extended bone loss on imaging to the middle or top third of the root. Periodontitis results in the loss of less than or equal to four teeth.

Exclusion Criteria:

* systemic illnesses
* pregnancy or lactation
* systemic antibiotics taken within the previous 6 months
* use of cholesterol reduction medication during the past 6 months
* subgingival scaling and root planing or surgical periodontal therapy in the last year
* chewing smokeless tobacco, smoking pipes or cigars 1 or more times per week, or smoking more than 20 cigarettes per week (1 pack per week) in the past 6 months

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People in Southern China
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
monocyte chemotactic protein-1，MCP-1 | Before surgery
  Concentration of MCP-1 in gingival crevicular fluids
monocyte chemotactic protein-1，MCP-1 | 1 month after surgery
  Concentration of MCP-1 in gingival crevicular fluids
monocyte chemotactic protein-1，MCP-1 | 3 months after surgery
  Concentration of MCP-1 in gingival crevicular fluids
oxidized low-density lipoprotein cholesterol, oxLDL | Before surgery
  Concentration of oxLDL in gingival crevicular fluids and serum
oxidized low-density lipoprotein cholesterol, oxLDL | 1 month after surgery
  Concentration of oxLDL in gingival crevicular fluids and serum
oxidized low-density lipoprotein cholesterol, oxLDL | 3 months after surgery
  Concentration of oxLDL in gingival crevicular fluids and serum

SECONDARY OUTCOMES:
interleukin-8，IL-8 | Before surgery
  Concentration of IL-8 in gingival crevicular fluids
interleukin-8，IL-8 | 1 month after surgery
  Concentration of IL-8 in gingival crevicular fluids
interleukin-8，IL-8 | 3 months after surgery
  Concentration of IL-8 in gingival crevicular fluids
triglycerides，TG | Before surgery
  Concentration of TG in serum
triglycerides，TG | 1 month after surgery
  Concentration of TG in serum
triglycerides，TG | 3 months after surgery
  Concentration of TG in serum
low-density lipoprotein cholesterol，LDL-C | Before surgery
  Concentration of LDL-C in serum
low-density lipoprotein cholesterol，LDL-C | 1 month after surgery
  Concentration of LDL-C in serum
low-density lipoprotein cholesterol，LDL-C | 3 months after surgery
  Concentration of LDL-C in serum
high-density lipoprotein cholesterol，HDL-C | Before surgery
  Concentration of HDL-C in serum
high-density lipoprotein cholesterol，HDL-C | 1 month after surgery
  Concentration of HDL-C in serum
high-density lipoprotein cholesterol，HDL-C | 3 months after surgery
  Concentration of HDL-C in serum
probing depth，PD | Before surgery
  The distance (mm) from the bottom of the periodontal pocket to the gingival margin was measured with a periodontal probe (UNC-15, Hu-Friedy, Chicago, IL) parallel to the long axis of the tooth. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth.
probing depth，PD | 1 month after surgery
  The distance (mm) from the bottom of the periodontal pocket to the gingival margin was measured with a periodontal probe (UNC-15, Hu-Friedy, Chicago, IL) parallel to the long axis of the tooth. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth.
probing depth，PD | 3 months after surgery
  The distance (mm) from the bottom of the periodontal pocket to the gingival margin was measured with a periodontal probe (UNC-15, Hu-Friedy, Chicago, IL) parallel to the long axis of the tooth. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth.
clinical attachment level，CAL | Before surgery
  The periodontal probe measures the distance (mm) from the bottom of the gingival sulcus or the bottom of the periodontal pocket to the cementoenamel boundary. The mesial, median and distal 6 points of the labial (buccal) and lingual surfaces were recorded for each tooth.
clinical attachment level，CAL | 1 month after surgery
  The periodontal probe measures the distance (mm) from the bottom of the gingival sulcus or the bottom of the periodontal pocket to the cementoenamel boundary. The mesial, median and distal 6 points of the labial (buccal) and lingual surfaces were recorded for each tooth.
clinical attachment level，CAL | 3 months after surgery
  The periodontal probe measures the distance (mm) from the bottom of the gingival sulcus or the bottom of the periodontal pocket to the cementoenamel boundary. The mesial, median and distal 6 points of the labial (buccal) and lingual surfaces were recorded for each tooth.
percentage of bleeding on probing，BOP% | Before surgery
  Gently probe to the bottom of the bag or gingival sulcus, take out the probe and observe for 10-15 seconds to see if there is any bleeding. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth. Calculate the percentage of bleeding sites.
percentage of bleeding on probing，BOP% | 1 month after surgery
  Gently probe to the bottom of the bag or gingival sulcus, take out the probe and observe for 10-15 seconds to see if there is any bleeding. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth. Calculate the percentage of bleeding sites.
percentage of bleeding on probing，BOP% | 3 months after surgery
  Gently probe to the bottom of the bag or gingival sulcus, take out the probe and observe for 10-15 seconds to see if there is any bleeding. The mesial, median and distal 6 sites of the labial (buccal) and lingual surfaces were recorded for each tooth. Calculate the percentage of bleeding sites.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China